CLINICAL TRIAL: NCT06872424
Title: The Effect of Psychosocial Skills Focused Group Psychoeducation on Functional Improvement, Treatment Compliance and Mental Well-Being in Schizophrenia Patients: a Randomised Controlled Study
Brief Title: The Effect of Psychosocial Skills Focused Group Psychoeducation in Schizophrenia Patients
Acronym: Schizophrenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Elif Güzide Emirza, Dr. Research Assistant, Gazi University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EGUEM
Record Dates: First submitted 2025-02-27; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia Patients; Psychoeducation; Functional Status; Treatment Outcome; Mental Development
Keywords: Schizophrenia; Psychoeducation; Functional recovery; Treatment adherence; Mental well-being
MeSH Terms: conditions — Schizophrenia; Treatment Adherence and Compliance; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Pre-test post-test control group study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effect of psychoeducation on schizophrenia patients (Experimental): Experimental and control group
  Interventions: Behavioral: psychosocial skills-oriented group psychoeducation

INTERVENTIONS:
Behavioral: psychosocial skills-oriented group psychoeducation — A 5-session Psychosocial Skills Focused Group Psychoeducation will be implemented, each session lasting approximately 60-90 minutes. In order to make the training more active and effective, the experimental group will be divided into small groups and divided into 3 groups and each group will be given 5 sessions of Psychosocial Skills Focused Group Psychoeducation once a week.

SUMMARY:
The aim of this study was to evaluate the effect of psychosocial skills-oriented group psychoeducation on functional recovery, treatment adherence and mental well-being in patients with schizophrenia. This research will be conducted in Giresun Community Mental Health Center. The study was planned as a randomized controlled pretest-posttest design. In addition to the Sociodemographic Information Form prepared by the researchers, the Functional Recovery Scale in Schizophrenia, the Modified Morisky Treatment Adherence Scale and the Warwick-Edinburgh Mental Well-Being Scale will be used to collect the data. The sample size was calculated as 34 people (experimental group= 17, control group= 17). Forms and scales will be applied to the experimental and control groups before psychoeducation and scales will be applied again to both groups after psychoeducation.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of psychosocial skills-oriented group psychoeducation on functional recovery, treatment adherence and mental well-being in patients with schizophrenia. This research will be conducted in Giresun Community Mental Health Center. The study was planned as a randomized controlled pretest-posttest design. In addition to the Sociodemographic Information Form prepared by the researchers, the Functional Recovery Scale in Schizophrenia, the Modified Morisky Treatment Adherence Scale and the Warwick-Edinburgh Mental Well-Being Scale will be used to collect the data. The sample size was calculated as 34 people (experimental group= 17, control group= 17). Forms and scales will be applied to the experimental and control groups before psychoeducation and scales will be applied again to both groups after psychoeducation. Forms and scales will be applied to the experimental and control groups before psychoeducation and scales will be applied again to both groups after psychoeducation. Thus, the effect of the psychoeducation program on the determined parameters will be evaluated. After the completion of the research, short-term counseling services will be provided to the control group in line with ethical principles. SPSS 25 package program will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Having a diagnosis of schizophrenia according to DSM-5 diagnostic criteria
2. To have continuity in the Community Mental Health Center
3. Being in remission (period without psychotic exacerbation) as a result of the evaluation of the outpatient clinic doctor,
4. To be mentally capable of understanding the questions posed
5. To have the cognitive competence to understand the training provided
6. Not having any visual or auditory disability
7. Graduating from at least primary school

Exclusion Criteria:

1. Refusing to participate in the study
2. Being under 18 years of age
3. Being illiterate in Turkish
4. Having Mental Retardation

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Functional Recovery Scale in Schizophrenia | 1 day
  Functional Recovery Scale: The scale is 5-point Likert-type and consists of 19 items. The maximum score that can be obtained from the scale is 95 and the minimum score is 19. Patients who score below 58 points are considered to have a low level of Functional Recovery, patients who score between 59-65 points are considered to have a moderate level of Functional Recovery, and patients who score 66 points and above are considered to have a high level.
Morisky Treatment Adherence Scale | 1 day
  Morisky Treatment Adherence Scale: The scale consists of 4 closed-ended questions with two options (yes/no). Medication adherence is assessed as high if "no" is answered to all questions (4 points), moderate if "yes" is answered to one or two questions (2-3 points), and low if "yes" is answered to three or four questions (0-1 pn).
Warwick-Edinburgh Mental Well-Being Scale | 1 day
  Warwick-Edinburgh Mental Well-Being Scale: The scale consists of 14 items and each question is scored between 1-5. The total score range is 14-70. A higher score indicates a higher level of mental well-being.

IPD SHARING:
Plan to Share IPD: No